CLINICAL TRIAL: NCT01447719
Title: Autopsy Follow-up of Subjects Previously Imaged With Florbetapir F 18 (18F-AV-45) PET in Trial 18F-AV-45-A07
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18F-AV-45-A16
Record Dates: First submitted 2011-05-20; First posted 2011-10-06 (Estimated); Results first posted 2012-05-07 (Estimated); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — florbetapir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: florbetapir F 18 — No study drug administered in this trial. Study subjects previously dosed with 18F-AV-45 in study 18F-AV-45-A07 (NCT00857415) are followed to autopsy in this extension study.
  Other Names: 18F-AV-45; Amyvid; florbetapir

SUMMARY:
This study is designed to test the relationship between measurements of brain amyloid using florbetapir F 18 PET imaging and true levels of amyloid plaque density as measured by histopathological assessment. The study will address the following specific aims:

1. To expand the number of subjects included in the A07 (NCT00857415) trial correlation analysis (measuring the correlation between the global visual rating of brain amyloid plaque density on an independent blinded read of the florbetapir F 18 PET scan and the cortical amyloid plaque density at autopsy as assessed by histopathology for subjects in the autopsy cohort).
2. To determine the sensitivity and specificity of an independent blinded visual read assessment of the florbetapir F 18 PET scan (Aβ+ or Aβ-) versus the final blinded neuropathological assessment made at autopsy.

ELIGIBILITY:
Inclusion Criteria:

Subjects are enrolled in this study if they:

* Met entrance criteria and were enrolled and imaged in trial 18F-AV-45-A07 (NCT00857415)
* Gave informed consent for the 18F-AV-45-A07 (NCT00857415) study procedures and brain donation consistent with the legal requirements of the State in which they are enrolled and the State in which they die
* Consent to participate in the 18F-AV-45-A16 (NCT01447719) extension protocol, if required by the IRB
* Reconfirm their consent to a research brain autopsy, if required by the IRB.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2010-03; Primary Completion 2011-03 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Research Site, Phoenix, Arizona
  - Research Site, Sun City, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Irvine, California
  - Research Site, Fort Myers, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Beach, Florida
  - Research Site, Miami Springs, Florida
  - Research Site, Orlando, Florida
  - Research Site, Sarasota, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Baltimore, Maryland
  - Research Site, Hattiesburg, Mississippi
  - Research Site, St Louis, Missouri
  - Research Site, Albany, New York
  - Research Site, New Hyde Park, New York
  - Research Site, Durham, North Carolina
  - Research Site, Centerville, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Charleston, South Carolina
  - Research Site, Johnson City, Tennessee

REFERENCES:
- [Derived] Clark CM, Pontecorvo MJ, Beach TG, Bedell BJ, Coleman RE, Doraiswamy PM, Fleisher AS, Reiman EM, Sabbagh MN, Sadowsky CH, Schneider JA, Arora A, Carpenter AP, Flitter ML, Joshi AD, Krautkramer MJ, Lu M, Mintun MA, Skovronsky DM; AV-45-A16 Study Group. Cerebral PET with florbetapir compared with neuropathology at autopsy for detection of neuritic amyloid-beta plaques: a prospective cohort study. Lancet Neurol. 2012 Aug;11(8):669-78. doi: 10.1016/S1474-4422(12)70142-4. Epub 2012 Jun 28. Erratum In: Lancet Neurol. 2012 Aug;11(8):658. PMID 22749065

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Demographic results are only provided for primary analysis populations of subjects who came to autopsy. Demographic characteristics for the entire population of 152 subjects are reported with the results of study A07 (NCT00857415).
Groups:
- Autopsy Cohort: End-of-life subjects consenting to brain donation at autopsy. Subjects received a single intravenous injection of 370 MBq florbetapir followed by a 10-minute PET scan 50 minutes post-injection.
Period: Overall Study
Arm/Group | Autopsy Cohort
Started | 152
Valid AV-45 Scan Acquired | 147
Deceased <2 Years After AV-45 Scan | 66
Completed | 59
Not Completed | 93
Not completed — Image acquisition failure | 2
Not completed — Invalid image or not imaged | 3
Not completed — Subject still living at end of study | 79
Not completed — Withdrawal by Subject | 2
Not completed — Family withdrew autopsy consent | 7

BASELINE CHARACTERISTICS:
Groups:
- All Autopsy Population: Group of subjects with valid images who came to autopsy within 2 years of scan
Arm/Group | All Autopsy Population
Number analyzed (Participants) | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.4 (12.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 29
Region of Enrollment [Number; unit: participants]
  United States | 59
Baseline clinical diagnosis [Number; unit: participants]
  AD diagnosis | 29
  Other dementing disorder | 13
  No history of cognitive impairment | 12
  Mild cognitive impairment | 5

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity Analysis in All Autopsy Population
Description: Sensitivity of florbetapir-PET scan to detect moderate to frequent amyloid plaques. Plaque density was calculated using CERAD (Consortium to Establish a Registry for AD) criteria. Florbetpir-PET scans were read by five independent readers blinded to clinical information using the binary read method (amyloid positive/negative).
Time Frame: at autopsy within 24 months of florbetapir PET scan
Population: 39 of 59 subjects from all autopsy population had moderate to frequent neuritic plaques at autopsy
Measure: Number; unit: participants
Groups:
- Subjects With Moderate or Frequent Plaques at Autopsy: Group of subjects with valid images who came to autopsy within 2 years of scan and had moderate to frequent neuritic plaques at autopsy (probable AD or definite AD)
Arm/Group | Subjects With Moderate or Frequent Plaques at Autopsy
Number analyzed (Participants) | 39
participants
  Florbetapir PET positive (majority interpretation) | 36
  Florbetapir PET negative (majority interpretation) | 3
Statistical Analysis 1: Comparison: Subjects With Moderate or Frequent Plaques at Autopsy; Proportion of subjects who had a positive scan based on majority of 5 blinded readers; Test type: Superiority or Other; Sensitivity = 92, 95% CI 2-sided [78 to 98] — 95% CI calculated by Wilson score method

2. Primary Outcome: Specificity Analysis in All Autopsy Population
Description: Specificity of florbetapir-PET scan to detect moderate to frequent amyloid plaques. Plaque density was calculated using CERAD criteria. Florbetpir-PET scans were read by five independent readers blinded to clinical information using the binary read method (amyloid positive/negative).
Time Frame: at autopsy within 24 months of florbetapir PET scan
Population: 20 of 59 subjects from the all autopsy population had no or sparse neuritic plaques at autopsy
Measure: Number; unit: participants
Groups:
- Subjects With no or Sparse Plaques at Autopsy: Group of subjects with valid images who came to autopsy within 2 years of scan and had no or sparse neuritic plaques at autopsy (no AD or possible AD)
Arm/Group | Subjects With no or Sparse Plaques at Autopsy
Number analyzed (Participants) | 20
participants
  Florbetapir PET positive (majority interpretation) | 0
  Florbetapir PET negative (majority interpretation) | 20
Statistical Analysis 1: Comparison: Subjects With no or Sparse Plaques at Autopsy; Proportion of subjects who had a negative scan based on majority of 5 blinded readers; Test type: Superiority or Other; Specificity = 100, 95% CI 2-sided [80 to 100] — 95% CI calculated by Wilson score method

3. Primary Outcome: Correlation of Florbetapir-PET Image and Amyloid Plaque Density
Description: Spearman's rank order correlation of the median visual read of the florbetapir-PET image and the amyloid plaque density assessed post-mortem by quantitative immunohistochemistry (IHC) averaged across 6 brain regions (precuneus, parietal cortex, frontal cortex, temporal cortex, posterior cingulate, anterior cingulate). Spearman's rank order correlation ranges from -1 to +1. A value of -1 indicates perfect negative correlation, and a value of +1 indicates a perfect positive correlation.
Time Frame: at autopsy within 24 months of florbetapir PET scan
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Arm/Group | All Autopsy Population
Number analyzed (Participants) | 59
Correlation coefficient | 0.76 [0.62 to 0.85]
Statistical Analysis 1: Comparison: All Autopsy Population; Spearman's Rank Order Correlation of the median semiquantitative read (three readers) and the quantitative IHC measurement of cortical amyloid plaque density averaged across six brain regions; Test type: Superiority or Other; p < 0.0001, Spearman's Rank Order Correlation test — A one-sided test (rho > 0) was performed with a significance level of alpha=0.05 to assess a significant correlation; Asymptotic standard error and 95 percent CI used Fisher z-transformation; Correlation coefficient = 0.76, 95% CI 2-sided [0.62 to 0.85], Standard Error of Mean 0.133

4. Secondary Outcome: Sensitivity Analysis in Subjects With Autopsy Within 1 Year of Scan
Description: Sensitivity of florbetapir-PET scan to detect moderate to frequent amyloid plaques. Plaque density was calculated using CERAD criteria. Florbetpir-PET scans were read by five independent readers blinded to clinical information using the binary read method (amyloid positive/negative).
Time Frame: at autopsy within 12 months of florbetapir PET scan
Population: 28 of 46 subjects who died within 1 year of scan had moderate to frequent neuritic plaques at autopsy
Measure: Number; unit: participants
Groups:
- Subjects With Moderate or Frequent Plaques at Autopsy: Group of subjects with valid images who came to autopsy within 1 years of scan and had moderate to frequent neuritic plaques at autopsy (probable AD or definite AD)
Arm/Group | Subjects With Moderate or Frequent Plaques at Autopsy
Number analyzed (Participants) | 28
participants
  Florbetapir PET positive (majority interpretation) | 27
  Florbetapir PET negative (majority interpretation) | 1
Statistical Analysis 1: Comparison: Subjects With Moderate or Frequent Plaques at Autopsy; Proportion of subjects who had a positive scan based on majority of 5 blinded readers; Test type: Superiority or Other; Sensitivity = 96, 95% CI 2-sided [80 to 100]

5. Secondary Outcome: Specificity Analysis in Subjects With Autopsy Within 1 Year of Scan
Description: as for outcome 2
Time Frame: at autopsy within 12 months of florbetapir PET scan
Population: 18 of 46 subjects who died within 1 year of scan had no or sparse neuritic plaques at autopsy
Measure: Number; unit: participants
Groups:
- Subjects With no or Sparse Plaques at Autopsy: Group of subjects with valid images who came to autopsy within 1 year of scan and had no or sparse neuritic plaques at autopsy (no AD or possible AD)
Arm/Group | Subjects With no or Sparse Plaques at Autopsy
Number analyzed (Participants) | 18
participants
  Florbetapir PET positive (majority interpretation) | 0
  Florbetapir PET negative (majority interpretation) | 18
Statistical Analysis 1: Comparison: Subjects With no or Sparse Plaques at Autopsy; Proportion of subjects who had a negative scan based on majority of 5 blinded readers; Test type: Superiority or Other; Specificity = 100, 95% CI 2-sided [78 to 100]

6. Other Pre Specified Outcome: Median Sensitivity and Specificity vs. CERAD Diagnosis
Description: Median sensitivity and specificity for 5 independent readers to detect moderate to frequent amyloid plaques (per CERAD criteria).
Time Frame: at autopsy within 24 months of florbetapir PET scan
Measure: Median (Full Range); unit: percentage of true positives/negatives
Arm/Group | All Autopsy Population
Number analyzed (Participants) | 59
percentage of true positives/negatives
  Sensitivity | 92 [69 to 95]
  Specificity | 95 [90 to 100]

7. Other Pre Specified Outcome: Individual Reader Results (All Scans With Autopsy)
Description: Reader results (number of false negatives and number of false positives) for blinded independent readers. There were a total of 39 positive and 20 negative scans based on histopathology at autopsy.
Time Frame: at autopsy within 24 months of florbetapir PET scan
Measure: Number; unit: florbetapir PET scans
Arm/Group | All Autopsy Population
Number analyzed (Participants) | 59
florbetapir PET scans
  Reader 1 - False Negatives | 3
  Reader 1 - False Positives | 1
  Reader 2 - False Negatives | 2
  Reader 2 - False Positives | 1
  Reader 3 - False Negatives | 5
  Reader 3 - False Positives | 1
  Reader 4 - False Negatives | 3
  Reader 4 - False Positives | 0
  Reader 5 - False Negatives | 12
  Reader 5 - False Positives | 2

8. Other Pre Specified Outcome: Individual Reader Results (Autopsy Within 1 Year of Scan)
Description: Reader results (number of false negatives and number of false positives) for blinded independent readers. There were a total of 28 positive and 18 negative scans based on histopathology at autopsy.
Time Frame: at autopsy within 12 months of florbetapir PET scan
Population: Includes only those subjects with time from scan to autopsy less than one year.
Measure: Number; unit: florbetapir PET scans
Groups:
- Autopsy Within 1 Year of Scan: Group of subjects with valid images who came to autopsy within 1 year of scan
Arm/Group | Autopsy Within 1 Year of Scan
Number analyzed (Participants) | 46
florbetapir PET scans
  Reader 1 - False Negatives | 1
  Reader 1 - False Positives | 1
  Reader 2 - False Negatives | 0
  Reader 2 - False Positives | 1
  Reader 3 - False Negatives | 3
  Reader 3 - False Positives | 0
  Reader 4 - False Negatives | 1
  Reader 4 - False Positives | 0
  Reader 5 - False Negatives | 7
  Reader 5 - False Positives | 2

ADVERSE EVENTS:
Time Frame: No adverse events were collected in this study, as this study only followed study A07(NCT01447719) subjects to autopsy. Adverse events are reported with study A07 (NCT00857415).
Description: No adverse events were collected in this study, as this study only followed study A07(NCT01447719) subjects to autopsy. Adverse events are reported with study A07 (NCT00857415).
Arm/Group | Autopsy Cohort
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days